CLINICAL TRIAL: NCT02184208
Title: Retrospective Review of Mechanically Ventilated Patients
Brief Title: Retrospective Review of Mechanically Ventilated Patients Using a Continuous Data Collection System.
Acronym: T3
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Brian Walsh, Research Coordinator / Research Associate, Boston Children's Hospital
Other Study IDs: IRB-P000011819
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Mechanical Ventilation; Acute Respiratory Distress Syndrome; Hypoxic Respiratory Failure
Keywords: ARDS; ALI; mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Device utlization following extubation
- Pulmonary mechanics

SUMMARY:
Today, the electronic medical record, microprocessor mechanical ventilators, and physiologic monitoring are under-utilized when translating research into decision support. Current medical informatic capabilities can be leveraged to calculate trends in measured parameters to initiate a paradigm shift in critical care from reaction-based treatment to proactive and plausibly preventative care. Therefore, the purpose of this study is to develop baseline understanding of our practice and how data collection utilizing a newly implemented system called T3. We would like to retrospectively review mechanically ventilated patients in which we have collected continuous data to test a newly developed analytic platform. Additionally we would like to compare these results to our standards of practice established by clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection will be determined by available data collected in the T3 system. We estimate 50 patients in which mechanical ventilator data has been collected utilizing the limited intellibridge modules (4 systems currently available to collect ventilator data).

Exclusion Criteria:

* Patient not connected to T3 data collection system.

Ages: 1 Day to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All mechanically ventilated patients in our medical surgical ICU.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Castineira D, Schlosser KR, Geva A, Rahmani AR, Fiore G, Walsh BK, Smallwood CD, Arnold JH, Santillana M. Adding Continuous Vital Sign Information to Static Clinical Data Improves the Prediction of Length of Stay After Intubation: A Data-Driven Machine Learning Approach. Respir Care. 2020 Sep;65(9):1367-1377. doi: 10.4187/respcare.07561. PMID 32879034
- [Derived] Walsh BK, Smallwood C, Rettig J, Kacmarek RM, Thompson J, Arnold JH. Daily Goals Formulation and Enhanced Visualization of Mechanical Ventilation Variance Improves Mechanical Ventilation Score. Respir Care. 2017 Mar;62(3):268-278. doi: 10.4187/respcare.04873. Epub 2017 Jan 10. PMID 28073993
- [Derived] Walsh BK, Smallwood CD, Rettig JS, Thompson JE, Kacmarek RM, Arnold JH. Categorization in Mechanically Ventilated Pediatric Subjects: A Proposed Method to Improve Quality. Respir Care. 2016 Sep;61(9):1168-78. doi: 10.4187/respcare.04723. Epub 2016 Jun 14. PMID 27303050

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Categorization: We retrospectively categorized the ventilation and oxygenation statuses of patients within our PICU utilizing 15 rules based algorithms. Targets were predetermined based on generally accepted practices. All patient categories were calculated and presented as a percent score (0-100%) of acceptable ventilation, acceptable oxygenation, barotrauma free and volutrauma free states.
Period: Overall Study
Arm/Group | Patient Categorization
Started | 278
Completed | 222
Not Completed | 56

BASELINE CHARACTERISTICS:
Arm/Group | Patient Categorization
Number analyzed (Participants) | 222
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3 [0.7 to 12.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 120
  More than one race | 33
  Unknown or Not Reported | 42
Region of Enrollment [Number; unit: participants]
  United States | 222

OUTCOME MEASURES:

1. Primary Outcome: Successful Extubation
Description: Successful extubation without the use of noninvasive ventilation or requiring reintubation
Time Frame: Within 24 hours of extubation
Measure: Count of Participants; unit: Participants
Groups:
- Device Utlization Following Extubation: The ERT score predicted device utilization
- Pulmonary Mechanics: Heart rate (HR), respiratory rate (RR), spontaneous respiratory rate (Spont. RR) and modified ventilation index (MVI) subcategory.
Arm/Group | Device Utlization Following Extubation | Pulmonary Mechanics
Number analyzed (Participants) | 104 | 222
Participants | 58 | 222

ADVERSE EVENTS:
Time Frame: Duration of ICU stay.
Groups:
- Device Utlization Following Extubation: Patients who were extubated were evaluated.
- Pulmonary Mechanics: All patients on mechanical ventilation were evaluated.
Arm/Group | Device Utlization Following Extubation | Pulmonary Mechanics
All-Cause Mortality (participants affected / at risk) | 9/104 | 20/222
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/222
Other Adverse Events (participants affected / at risk) | 0/104 | 0/222

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes